CLINICAL TRIAL: NCT01495247
Title: A Dose-finding Phase Ib Study Followed by an Open-label, Randomized Phase II Study of BEZ235 Plus Paclitaxel in Patients With HER2 Negative, Inoperable Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase Ib/II Trial of BEZ235 With Paclitaxel in Patients With HER2 Negative, Locally Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study did not meet Phase Ib primary objective to establish the maximum tolerated dose/recommended dose for Phase II
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235B2101; 2011-002400-32 (EudraCT Number)
Record Dates: First submitted 2011-09-30; First posted 2011-12-19 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-09

CONDITIONS: Inoperable Locally Advanced Breast Cancer; Metastatic Breast Cancer (MBC)
Keywords: Locally advanced; metastatic; breast cancer; HER2 negative; PI3K pathway; paclitaxel; mTOR inhibitor
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — dactolisib; Paclitaxel

ARMS (2):
- BEZ235 100 mg bid + paclitaxel 80 mg (phase lb) (Experimental): Increasing doses of oral BEZ235 100 mg administered on a continuous twice daily (BID) schedule + weekly paclitaxel infusion at a fixed dose of 80 mg/m2. Treatment was organized into cycles of 28 days.
  Interventions: Drug: BEZ235; Drug: Paclitaxel
- BEZ235 200 mg bid + paclitaxel 80 mg (phase lb) (Experimental): Increasing doses of oral BEZ235 200 mg administered on a continuous twice daily (BID) schedule + weekly paclitaxel infusion at a fixed dose of 80 mg/m2. Treatment was organized into cycles of 28 days
  Interventions: Drug: BEZ235; Drug: Paclitaxel

INTERVENTIONS:
Drug: BEZ235 — Doses of oral BEZ235 (BID), supplied as 50mg, 200mg, 300mg or 400mg in SDS sachets, together with standard weekly paclitaxel at a fixed dose (80mg/m²) during 1h by i.v. in infusion.
Drug: Paclitaxel — The paclitaxel infusion will be given in the morning and directly thereafter the BEZ235 dose will be given.
  BEZ235 doses will be escalated in cohorts of 3 to 6 patients guided by an adaptive Bayesian logistic regression model with overdose control until MTD/RP2D has been established. The initial dose level for the first cohort will be 200mg (BID), and then based on the Bayesian model the dose may be escalated to 300mg, 400mg, 500mg or 600mg for the next cohorts.

SUMMARY:
This is a prospective, multi-center, open-label, phase Ib/ II study (two parts) with patients that have locally advanced or metastatic HER2 negative breast cancer. The first part (phase Ib) will investigate the MTD / Recommended Phase 2 Dose (RP2D) of the combination therapy of BEZ235 twice daily (b.i.d.) and weekly paclitaxel using a Bayesian model. When MTD/ RP2D is established the second part (phase II) will start. Phase II will evaluate the efficacy and the safety of weekly paclitaxel alone compared to weekly paclitaxel plus BEZ235 bid.

ELIGIBILITY:
Inclusion Criteria (phase lb):

* Females with Breast cancer that is histologically or cytologically confirmed, HER2 negative and locally advanced or metastatic as confirmed by radiology
* ECOG performance status 0 and 1
* Adequate bone marrow and organ function

Exclusion Criteria (Phase lb):

* Previous treatment with PI3K and/or mTOR inhibitors
* Symptomatic Central Nervous System (CNS) metastases
* Concurrent malignancy or malignancy in the last 5 years prior to start of study treatment
* Wide field radiotherapy ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to starting study drug
* Active cardiac disease (e.g. LVEF less than institutional lower limit of normal, QTcF > 480 msec, unstable angina pectoris, ventricular, supraventricular or nodal arrhythmias)
* Inadequately controlled hypertension
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BEZ235 and/or paclitaxel
* Treatment at start of study treatment with drugs with a known risk to induce Torsades de Pointes, moderate and strong inhibitors or inducers of isoenzyme CYP3A4, warfarin and coumadin analogues, LHRH agonists
* Sensitivity to paclitaxel treatment
* Uncontrolled diabetes mellitus
* Pregnant or nursing (lactating) woman

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2014-05-19 (Actual); Study Completion 2014-05-19 (Actual)

PRIMARY OUTCOMES:
Phase lb: Dose Limiting Toxicities (DLTs) the first cycle of treatment | At first treatment intake (Cycle 1 Day 1 = C1D1), C1D8, C1D15, C1D22 and C2D1 [a cycle = 4 weeks = 28 days]
  DLT is defined as treatment-related toxicity (classified according Common Toxicity Criteria for Adverse Events (CTCAE) Version 4) occurring during the first 28 treatment days and meeting specific protocol-predefined criteria.
  The information will be integrated in a Bayesian logistic regression model with overdose control to estimate the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Phase lb: Frequency and severity of adverse events | At screening, every week (C1D1, C1D8, C1D15, C1D22, C2D1, C2D8, etc.) until 30-45 days after treatment discontinuation [estimated time frame: 18 months].
  Incidence of adverse events (based on CTCAE Version 4) summarized by system organ class and/or preferred term, severity and relation to study treatment.
Phase lb: Progression free survival (PFS) | At first treatment intake, every 8 weeks (C3D1, C5D1, C7D1, etc.) until disease progression or death for any cause [estimated time frame: 18 months].
  PFS is defined as the time from start of treatment to objective tumor progression or death from any cause. Radiological assessments will be performed every 8 weeks.
Phase lb: Overall Response Rate (ORR) | At first treatment intake, every 8 weeks (C3D1, C5D1, C7D1, etc.) during the study [estimated time frame: 18 months].
  Proportion of patients with a best overall response of CR or PR according to RECIST 1.1
Phase lb: Clinical Benefit Rate (CBR) | At first treatment intake, every 8 weeks (C3D1, C5D1, C7D1, etc.) during the study [estimated time frame: 18 months].
  Proportion of patients with a best overall response of CR, PR or SD with a duration of 24 weeks or longer according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- France (2):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Saint-Herblain Cédex
- Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia, Spain

REFERENCES:
- See also: Results for CBEZ235B2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13703